CLINICAL TRIAL: NCT05011578
Title: Evaluation of Long-term Clinical and Radiographic Outcomes of Radio-capitellar Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rad-Hop
Record Dates: First submitted 2021-08-09; First posted 2021-08-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Radiocapitellar Dislocation
Keywords: radio-capitellar fracture; interventional study; Radiographic assessment; radio-capitellar prosthetic arthroplasty; long term clinical results; long term radiographic results; radio-capitellar prosthesis; radiographic results; clinical results

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- clinical and radiographic findings after surgical treatment for radiocapitellar fracture (Experimental): 30 patients will be included in a interventional study for an evaluation of the clinical and radiographic finding after at least 10 years after radiocapitellar surgery
  Interventions: Radiation: Radiographic assessment

INTERVENTIONS:
Radiation: Radiographic assessment — Radiographic assessment after at least 10 years after radiocapitellar surgical treatment

SUMMARY:
The aim of this study is to collect clinical and radiographic data from the case histories of patients surgically treated for radio-capitellar fracture and undergoing prosthetic replacement with a modular metal radio-capitellar prosthesis with smooth stem at the Shoulder-Elbow Department of the Rizzoli Orthopaedic Institute, in order to evaluate the clinical and radiographic results at least 10 years after surgery.

DETAILED DESCRIPTION:
The aim of the study is to collect clinical and radiographic data from the case history of patients (about 30 cases) surgically treated from 2003 to 2011 at the Shoulder-Elbow Department of the Rizzoli Orthopaedic Institute for radio-capitellar fracture with prosthetic replacement with a modular metal radio-capitellar prosthesis with smooth stem in order to evaluate the clinical and radiographic results at least 10 years after treatment. Patients will be contacted to perform a clinical examination and radiographic control at the Rizzoli Orthopaedic Institute.

This is an interventional study with clinical and radiographic evaluation, at FU of at least 10 years, of patients treated surgically with prosthetic replacement for radio-capitellar fracture at the Shoulder-Elbow Department of the Rizzoli Orthopaedic Institute.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of radial capitate implantation surgery
2. Males and Females
3. Patients surgically treated for radial capitellum fracture undergoing prosthetic replacement with smooth-stemmed modular metal radial capitellum prosthesis at the Shoulder-Elbow Department of the Rizzoli Orthopaedic Institute from 2003 to 2011.

Exclusion Criteria:

1. < 18 years old at the time of surgery
2. Patients treated with radial capitellum prosthesis implantation in fracture outcomes (e.g., secondary instability)
3. Patients who at the time of telephone contact have contraindications to the execution of radiographic examination
4. All available patients will be invited to perform the clinical examination and radiographic examination. If some patients are unable to undergo radiography due to possible contraindications, they will still be seen to collect the primary clinical outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Mayo elbow performance score (MEPS): | At least 10 years after radiocapitellar prosthesis surgical treatment
  MEPS score assesses the presence of pain with a score of 0 to 45, Range of Motion with a score of 0 to 20, elbow stability with a score of 0 to 10, and the ability to perform 5 activities of daily living (combing, eating, personal hygiene, dressing, and putting on shoes) to each of which 5 points are assigned. It provides a result from 0 to 100 where results above 90 are defined as excellent, results between 75 and 89 are defined as good, between 60 and 74 are defined as sufficient and below 59 as poor.

SECONDARY OUTCOMES:
Broberg - Morrey Score | At least 10 years after radiocapitellar prosthesis surgical treatment
  The Broberg and Morrey assessment system is a 100-point system that summarizes data from the medical record, personal interview, and biomechanics laboratory examination. It consists of four sections: motion (40 points), strength (20 points), stability (5 points), and pain (35 points). In the final evaluation 95-100 points indicate an excellent result; 80-94 points, a good result; 60-79 points, a fair result; ≤60 points, a poor result. The result can be considered satisfactory if the outcome is rated as good or excellent and unsatisfactory if it is fair or poor.
Short Form-12 (SF-12): | At least 10 years after radiocapitellar prosthesis surgical treatment
  SF-12 serves as a generic indicator of quality of life and assesses the individual's subjective perception of health, understood as biopsychosocial well-being. Through 12 of the 36 questions of the original questionnaire, the SF-12 investigates 8 different aspects related to health status: physical activity, role limitations due to physical health, emotional state, physical pain, perception of general health status, vitality, social activities and mental health; the synthesis of the total scores allows to build two synthetic indices, a physical health index (PCS-12) and a mental health index (MCS-12). The lower the score of the two indices, indicatively below 20 points, the greater the level of disability.
Treatment opinion post- surgery | At least 10 years after radiocapitellar prosthesis surgical treatment
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial (24 months follow-up). All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".
Radiographic assesment (RX) | At least 10 years after radiocapitellar prosthesis surgical treatment
  Radiographic assessment is useful to document re-ruptures, mobilizations and calcifications of the interested site

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Marsh JP, Grewal R, Faber KJ, Drosdowech DS, Athwal GS, King GJ. Radial Head Fractures Treated with Modular Metallic Radial Head Replacement: Outcomes at a Mean Follow-up of Eight Years. J Bone Joint Surg Am. 2016 Apr 6;98(7):527-35. doi: 10.2106/JBJS.15.00128. PMID 27053580
- [Background] Morrey BF, Askew LJ, Chao EY. A biomechanical study of normal functional elbow motion. J Bone Joint Surg Am. 1981 Jul;63(6):872-7. PMID 7240327
- [Background] Lott A, Broder K, Goch A, Konda SR, Egol KA. Results after radial head arthroplasty in unstable fractures. J Shoulder Elbow Surg. 2018 Feb;27(2):270-275. doi: 10.1016/j.jse.2017.10.011. PMID 29332663
- [Background] Harrington IJ, Sekyi-Otu A, Barrington TW, Evans DC, Tuli V. The functional outcome with metallic radial head implants in the treatment of unstable elbow fractures: a long-term review. J Trauma. 2001 Jan;50(1):46-52. doi: 10.1097/00005373-200101000-00009. PMID 11231669
- [Background] Fowler JR, Goitz RJ. Radial head fractures: indications and outcomes for radial head arthroplasty. Orthop Clin North Am. 2013 Jul;44(3):425-31, x. doi: 10.1016/j.ocl.2013.03.013. Epub 2013 Apr 17. PMID 23827844